CLINICAL TRIAL: NCT00584324
Title: The Effect of Depth of Anesthesia on Implicit Memory
Brief Title: Depth of Anesthesia on Implicit Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB No: 12634
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Anesthesia, General; Memory
Keywords: elective surgery; general anesthesia; implicit memory
MeSH Terms: interventions — Consciousness Monitors; 61-bis(1-adamantylcarbamoyl)-1,2-methano(60)fullerene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bispectral Index (BIS) 40 (Experimental): Target BIS 40
  Interventions: Combination Product: BIS 40; Combination Product: BIS 60
- Bispectral Index (BIS) 60 (Experimental): Target BIS 60
  Interventions: Combination Product: BIS 40; Combination Product: BIS 60

INTERVENTIONS:
Combination Product: BIS 40 — Mini-mental state exam: For subjects > 60, this exam will be administered pre-operatively.
  Spielberger State-Trait anxiety test: Spielberger test just before being taken to the operating room.
  Spoken word-stem completion test: After discharge from recovery but within 24 hrs. post surgery, this test along with the anxiety test will be administered.
  Bispectral Index Monitor: The physiologic monitor is used intraoperatively to assess surgical anesthesia.
  Audio File: Playing an audio file (a list of spoken words) via headphones under general anesthesia during the surgical procedure.
  Other Names: Mini-mental state exam; Spielberger State-Trait anxiety test; Spoken word-stem completion test; Bispectral Index Monitor; Audio File
Combination Product: BIS 60 — Mini-mental state exam: For subjects > 60, this exam will be administered pre-operatively.
  Spielberger State-Trait anxiety test: Spielberger test just before being taken to the operating room.
  Spoken word-stem completion test: After discharge from recovery but within 24 hrs. post surgery, this test along with the anxiety test will be administered.
  Bispectral Index Monitor: The physiologic monitor is used intraoperatively to assess surgical anesthesia.
  Audio File: Playing an audio file (a list of spoken words) via headphones under general anesthesia during the surgical procedure.
  Other Names: Mini-mental state exam; Spielberger State-Trait anxiety test; Spoken word-stem completion test; Bispectral Index Monitor; Audio File

SUMMARY:
Purpose of this study is to see if different levels of anesthesia have an effect on hearing spoken words without awareness of having heard them or anxiety after surgery.

DETAILED DESCRIPTION:
Amnesia (lack of recall) is one of the most important goals of general anesthesia. Inadvertent free recall during a major surgical procedure is not only inhumane, but also predisposes the patient to morbidity such as post-traumatic stress disorder. Therefore, it is standard practice among anesthesiologists to inquire about free (explicit) recall during a post-anesthetic visit.

Free recall requires a functional long term memory. Historically, lack of free recall during general anesthesia has been regarded as complete absence of long term memory activity. However, recent evidence suggests that the relationship between general anesthesia and memory is more complex than previously thought.

Objectives of the proposed are twofold: (1) to test the presence of implicit memory under two different planes of surgical general anesthesia in elderly males (55-90 years old) during a uniform surgical procedure (urologic procedures via transurethral approach) (2) to compare the pre and postoperative anxiety levels as a marker of clinical significance of operational implicit memory function.

The study is divided into three phases: pre-operative, operative, and post-operative.

Pre-operative phase will consist of a cognitive function test (mini-mental state exam). This will be administered at the urology or pre-operative anesthesia clinic visit, after obtaining the informed consent of the patient.

Operative phase will start with a baseline anxiety test (Spielberger state-trait anxiety test) just before being taken to the operating room. This will be followed by playing an audio file (a list of spoken words) via headphones under general anesthesia during the surgical procedure.

Post-operative phase will have of a spoken word-stem completion test (just before discharge from the hospital) and a repeat of the anxiety test mentioned above (2 to 3 weeks post-operatively).

ELIGIBILITY:
Inclusion Criteria:

* Persons signing informed consent
* Elective general surgery for orthopedics (external or internal fixation) or urologic (transurethral)
* Literate
* Native English speaking

Exclusion Criteria:

* Hearing impaired
* History of cognitive dysfunction
* Subjects requiring post-operative sedation for any indication

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To test the presence of implicit memory under two different planes of surgical general anesthesia in patients undergoing urologic (transurethral) or orthopedic (internal and external fixation) procedures | 3 years

SECONDARY OUTCOMES:
To compare the pre and postoperative anxiety levels as a marker of clinical significance of operational implicit memory function. | 3

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet S. Ozcan, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No